CLINICAL TRIAL: NCT05350852
Title: To Evaluate the Safety, Efficacy and Pharmacokinetics of ThisCART19A in Patients With MRD Positive Acute B-cell Leukemia
Brief Title: Evaluate the Safety, Efficacy and Pharmacokinetics of ThisCART19A in Patients With MRD+ B-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, President/Proffessor, Zhejiang University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT400-005
Record Dates: First submitted 2022-04-09; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: B-ALL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ThisCART19A 5×10^6 cells/kg for dose level 1 (Experimental): Patients will receive 5×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- ThisCART19A 8×10^6 cells/kg for dose level 2 (Experimental): Patients will receive 8×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A
- ThisCART19A 12×10^6 cells/kg for dose level 3 (Experimental): Patients will receive 12×10^6 cells/kg of ThisCART19A
  Interventions: Biological: ThisCART19A

INTERVENTIONS:
Biological: ThisCART19A — ThisCART19A is a new type CAR-T cells therapy for patients with acute B-cell leukemia

SUMMARY:
This is an open label, phase I study to assess the safety, efficacy and pharmacokinetics of ThisCART19A in patients with MRD+ B-ALL

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. All subjects or legal representatives must sign a voluntary letter of consent approved by the IRB in person prior to the commencement of any screening procedure;
  2. Patients diagnosed with B-ALL according to the Chinese Guidelines for the Diagnosis and Treatment of Adult Acute Lymphoblastic Leukemia (2021 edition);
  3. There is no gender limitation, age 18-65 (upper limit not included);
  4. Disease status ≥CR2 with bone marrow flow cytometry MRD≥0.1%.
  5. Patients with Ph+ R/R ALL who failed after 2-line TKI treatment, were intolerant to TKI treatment or were not suitable for TKI treatment;
  6. The expected survival time is ≥12 weeks;
  7. ECOG score 0-1;
  8. Had good organic function during screening
  9. CD19 was still expressed on leukemia cells in bone marrow, peripheral blood or biopsy tissue by flow cytometry, results within one month prior to informed consent are acceptable (after the last treatment).

Exclusion Criteria:

1. Allergic to preconditioning measures.
2. Patients with other malignancies other than B-cell malignancies within 5 years prior to screening. Patients with cured skin squamous carcinoma,basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited.
3. Uncontrollable bacterial, fungal and viral infection during screening.
4. Patients had pulmonary embolism within 3 months prior to enrollment.
5. Had intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases prior to enrollment.
6. Imaging confirmed the presence of central nervous system involvement (both primary and secondary) and obvious symptoms at the time of screening.
7. < 100 days after hematopoietic stem cell transplantation.
8. Active HBV or HCV or HIV or Syphilis infection. HBV-DNA < 2000 IU/mL can be enrolled, but should admitted to use anti-virus drugs such as entecavir, tenufovir, etc, and supervisory the relative indication during the treatment.
9. Combined systemic steroid use (e.g., prednisone ≥20mg) within 3 days prior to screening. Or systemic diseases that require long-term use of immunization Inhibitor.
10. Vaccinated with influenza vaccine within 2 weeks prior to cleansing (SARS-COV19 can be included, inactivated, live/non-live adjuvant vaccinations allowed to be included) .
11. Patients who are receiving GvHD treatment; Patients without GvHD and who had stopped immunosuppressive drugs for at least 1 month were eligible for inclusion.
12. Women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after cell infusion. Male subjects who plan pregnancy within 1 year after infusion.
13. Any ineligibility conditions considered by the investigator that may increase the risk of the subject or interfere with the results of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after ThisCART19A infusion
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.
The incidence of all grade TEAEs and ≥3 grade TEAEs | Up to 2 years after ThisCART19A infusion
  Incidence of treatment-emergent adverse events (TEAEs) and ≥3 grade TEAEs

SECONDARY OUTCOMES:
Relapse-Free Survival | 24 months
  Defined as the time from the infusion of ThisCART19A cells to the occurrence of hematologic relapse or death from any cause.Hematologic recurrence was defined as ≥5% of bone marrow lymphoblasts or extramedullary recurrence after CR or CRi
MRD response rate | At Month 1, 2, 3
  Percentage of participants with minimal residual disease (MRD) response in patients with CR (complete response) and CRi (CR with incomplete blood count recovery) ; MRD Response is defined as leukemic cells in bone marrow <0.01% by flow cytometry (sensitivity at least 0.001%)
The change characteristics of chimeric antigen receptor(CAR)-T cell number and copy number in patients after infusion | 3 months
  Track CAR-T cells expansion in patients after infusion by flow cytometry and qPCR
Changes in cytokine level after ThisCART19A infusion. | 3 months
  Calculate the change of cytokine level in peripheral blood by flow cytometry after ThisCART19A infusion. Cytokines include IL-1β、IL-2、IL-4、IL-6、IL-8、IL-10、IL-12、IL-17、TNF-α、IFN-γ、TGF-β.
Changes in immune effect cells count after ThisCART19A infusion. | 3 months
  Calculate the change of immune effect cells count in peripheral blood by flow cytometry after ThisCART19A infusion. Immune effect cells include T cell, B cell, NK cell.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, Doctor, Principal Investigator — The first hospital affiliated Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China